CLINICAL TRIAL: NCT04194398
Title: OCS Lung Expand Post-Approval Study - Expand Follow-Up Data Collection
Status: Completed | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-LUN-122018
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: OCS Lung System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- OCS Expand Trial Cohort: All patients previously enrolled in the EXPAND Lung trial.
  Interventions: Device: OCS Lung System

INTERVENTIONS:
Device: OCS Lung System — Patients previously transplanted with lungs preserved on the OCS Lung System in the Expand Lung study.

SUMMARY:
Collection of five year follow-up data on patients who have already participated in the EXPAND Lung trial and have had transplants with donor lungs preserved on the OCS Lung System.

DETAILED DESCRIPTION:
The purpose of this continuation study is to collect five year follow-up data on patients who have already participated in the EXPAND Lung trial and have had transplants with donor lungs preserved on the OCS Lung System. The EXPAND Lung trial results have been presented and have shown positive results in the use of expanded criteria donor lungs and patient follow-up, post-transplant. The current study is being conducted to continue to collect follow-up on participants in the EXPAND study, in order to evaluate long-term patient survival status and BOS diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Registered male or female primary double lung transplant candidate
* Age ≥18 years old
* Signed: 1) written informed consent document and 2) authorization to use and disclose protected health information

Exclusion Criteria:

* Prior solid organ or bone marrow transplant
* Single lung recipient
* Chronic use of hemodialysis or diagnosis of chronic renal insufficiency

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients previously enrolled in the Expand Lung trial who received lungs preserved on the OCS Lung System.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Patient and graft survival | 2 years
  Survival of graft and survival as evaluated at follow-up visit/call with patient or health care provider.
Patient and graft survival | 3 years
  Survival of graft and survival as evaluated at follow-up visit/call with patient or health care provider.
Patient and graft survival | 4 years
  Survival of graft and survival as evaluated at follow-up visit/call with patient or health care provider.
Patient and graft survival | 5 years
  Survival of graft and survival as evaluated at follow-up visit/call with patient or health care provider.
Presence or absence of bronchiolitis obliterans sydrome (BOS) | 2 years
  Evaluation of BOS as determined by follow-up evaluation visit/call with patient or health care provider.
Presence or absence of bronchiolitis obliterans sydrome (BOS) | 3 years
  Evaluation of BOS as determined by follow-up evaluation visit/call with patient or health care provider.
Presence or absence of bronchiolitis obliterans sydrome (BOS) | 4 years
  Evaluation of BOS as determined by follow-up evaluation visit/call with patient or health care provider.
Presence or absence of bronchiolitis obliterans sydrome (BOS) | 5 years
  Evaluation of BOS as determined by follow-up evaluation visit/call with patient or health care provider.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California at Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
- Hospitals Leuven, Leuven, Belgium
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Loor G, Warnecke G, Villavicencio MA, Smith MA, Zhou X, Kukreja J, Ardehali A, Hartwig MG, Daneshmand MA, Hertz MI, Huddleston SJ, Haverich A, Madsen JC, Neyrinck A, Van Raemdonck D. Long-term outcomes of the international EXPAND trial of Organ Care System (OCS) Lung preservation for lung transplantation. EClinicalMedicine. 2025 Jul 8;85:103334. doi: 10.1016/j.eclinm.2025.103334. eCollection 2025 Jul. PMID 40686680